CLINICAL TRIAL: NCT01896167
Title: Study of Migraine With Aura Inducing Characteristics and Effects on the Cerebral Arteries by Hypoxia in a Humane Experimental Migraine Model
Brief Title: Migraine With Aura Inducing Characteristics and Effects on the Cerebral Arteries and Blood Flow by Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Nanna Arngrim, MD, medical doctors, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-4-2012-182
Record Dates: First submitted 2013-06-21; First posted 2013-07-11 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Headache; Migraine; Aura
Keywords: Headache; Migraine; Aura; Cerebral hemodynamics
MeSH Terms: conditions — Headache; Migraine Disorders; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypoxia (Active Comparator): Inhalation of air with 8-12% oxygen content
  Interventions: Other: Hypoxia
- Atmospheric air (Placebo Comparator): Inhalation of atmospheric air, with oxygen content at 21%
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Hypoxia — Inhalation of hypoxic air (8-12% oxygen content)
  Arms: Hypoxia
Other: Placebo — Inhalation of atmospheric air
  Arms: Atmospheric air

SUMMARY:
In this study the investigators will investigate the following hypothesis

* that hypoxia induce migraine headache and migraine aura
* the aura phase is associated with a spreading reduction in cerebral blood flow
* the migraine headache is associated with dilatation of intra- and extracerebral arteries
* the migraine headache is associated with changes in brain metabolism
* the pre-ictal stage of a migraine attack with aura is associated with specific patterns in neural activity.

DETAILED DESCRIPTION:
To investigate migraine with aura symptoms during and after hypoxia.

With magnetic resonance imaging the investigators will investigate changes in

* regional cerebral blood flow (rCBF)
* resting state functional connectivity
* circumference of the middle cerebral artery(MCA), internal carotic artery, superficial temporal artery, medial meningeal artery, external carotic artery
* brain metabolism

And compare these changes with a aged match healthy control group.

ELIGIBILITY:
Inclusion Criteria:

Migraine with aura patients and Helthy volunteers as controls:

* Aged 18-40
* 50-100 kg

Exclusion Criteria:

* Tension type headache more than 5 days/month
* Other primary headaches
* Daily medication except contraceptives
* Drug taken within 4 times the halflife for the specific drug except contraceptives
* Pregnant or lactating women
* Headache or migraine attack within the last 48 hours before start of trial
* Hypertension
* Hypotension
* Respiratory or cardiac disease
* smoking

Extra exclusion Criteria for healthy volunteers:

* migraine at present or earlier in life
* parents, sibling or children who suffer or have suffered from migraine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Headache and aura | 24 h
  Comparison between hypoxia and placebo (atmospheric air)

SECONDARY OUTCOMES:
artery circumference | Baseline, 120 and 200 min
  Hypoxia induced changes in intra- and extracranial circumference
Cerebral blood flow | Baseline, 120 and 200 min
  Hypoxia induced changes in cerebral blood flow
BOLD response in visual cortex | Baseline, 170 min and 220 min
  Hypoxia induced changes in BOLD response
Brain metabolism | Baseline, 180 min and 230 min post hypoxia
  Hypoxia induced changes in brain metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Arngrim, MD, Principal Investigator — Department of Neurology, Glostrup Hospital
Locations (1):
- Nanna Arngrim, Glostrup Municipality, Denmark